CLINICAL TRIAL: NCT02673632
Title: The Influence of Anti-Müllerian Hormone on Ovarian Responsiveness to Ovulation Induction With Gonadotrophins in Women With Polycystic Ovarian Syndrome
Brief Title: The Influence of AMH on Ovarian Responsiveness to Ovulation Induction With GnRH in Women With PCOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, Assistant professor, Ain Shams Maternity Hospital
Other Study IDs: ASU2016
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: Anti-Müllerian hormone; Ovarian stimulation; Polycystic ovary syndrome; Intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — hMG-IBSA; Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Merional ® — Using the long protocol of controlled ovarian hyperstimulation (COH). Down regulation by (Decapeptyl ®, Ferring) 0.1mg subcutaneously once daily starting from day 18 of the preceding cycle, human menopausal gonadotrophin (hMG) (Merional ®, IBSA) 75 IU starting from cycle day two after confirmation of down regulation (thin endometrium, number of follicular activity, E2 < 50 pg/mL). hMG dose is optimized according to age, BMI, antral follicles count (AFC), the local protocol, FSH level and previous response. Usually PCO patients start by 150 IU.
  Other Names: Decapeptyl ®

SUMMARY:
The investigator suggests that PCOS women with high AMH levels are resistant to ovarian stimulation and may need adjustment of the dose of gonadotrophin.

DETAILED DESCRIPTION:
There is a correlation between high levels of AMH and the severity of PCOS. Excessive AMH may have a negative effect on the sensitivity of the resting follicles to gonadotropins.

This is an observational prospective study to investigate the impact of circulating AMH on gonadotrophin induction in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women of age 18 - 35 years
* BMI 20 - 30 kg/m2
* Anovulatory infertility
* Diagnosis of PCOS based on Rotterdam consensus criteria (two of three criteria: Oligo/anovulation, hyperandrogenaemia and sonographic appearance of polycystic ovaries)

Exclusion Criteria:

* Women Above 35 years or under 18 years
* Women with BMI above 30 kg/m2 or under 20 kg/m2
* Normally ovulating women
* Patients with marked hyperandrogenaemia were screened for congenital adrenal hyperplasia (by measuring serum concentration of 17alpha hydroxyl-progesterone) or Patients with Cushing syndrome (by measuring urinary free cortisol)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population comprises women with PCOS, fulfilling the inclusion criteria, attending to Ain Shams University Maternity Hospital, assisted reproductive technology (ART) Unit, during the study period, who are planning for Intracytoplasmic sperm injection (ICSI).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Good response to hMG therapy defined as occurrence of > 3 mature follicles after treatment. | 30 days
  Good response to hMG therapy defined as occurrence of > 3 mature follicles after treatment.

REFERENCES:
- [Background] Amer SA, Mahran A, Abdelmaged A, El-Adawy AR, Eissa MK, Shaw RW. The influence of circulating anti-Mullerian hormone on ovarian responsiveness to ovulation induction with gonadotrophins in women with polycystic ovarian syndrome: a pilot study. Reprod Biol Endocrinol. 2013 Dec 17;11:115. doi: 10.1186/1477-7827-11-115. PMID 24341292